CLINICAL TRIAL: NCT01167764
Title: Effect of Tranexamic Acid on Prevention of Recurrence of Hemoptysis: Multicenter, Prospective, Randomized, Double-blind Phase 3 Trial
Brief Title: Effect of Tranexamic Acid on Prevention of Recurrence of Hemoptysis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Joon Yim / Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SNUH-tranexamic acid
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Hemoptysis
Keywords: hemoptysis; recurrence
MeSH Terms: conditions — Hemoptysis; Recurrence | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tranexamic acid (Active Comparator): tranexamic acid 250mg po 3 times/day for 1 months
  Interventions: Drug: tranexamic acid, placebo
- placebo (Placebo Comparator): placebo po 3 times/day for 1 months
  Interventions: Drug: tranexamic acid, placebo

INTERVENTIONS:
Drug: tranexamic acid, placebo — tranexamic acid 250mg tid for 1 months vs. placebo for 1 months

SUMMARY:
Hemoptysis is one of the serious complication of many pulmonary diseases. Upto now, there is no proven medical treatment in recurrence of hemoptysis. The investigators will conduct a randomized, placebo controlled trial of tranexamic acid, which can reduce the recurrence of hemoptysis.

ELIGIBILITY:
Inclusion Criteria:

* age: >=20 and <=75
* ER visit or admission for hemoptysis
* no evidence of hemoptysis on screening

Exclusion Criteria:

* anticoagulation treatment
* Cr >= 2.0 mg/dL or urinary protein >= 2+ or who received renal replacement treatment
* hepatic failure: total bilirubin >= 1.5 mg/dL or AST or ALT >= 1.5 of upper normal limit level
* hypersensitivity to tranexamic acid
* pregnant woman
* fertile female who don't use contraception

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
the proportion of recurrence of hemoptysis | 6 month: 1months medication + 5months observation

SECONDARY OUTCOMES:
time to recurrence | 6 month: 1months medication + 5months observation

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul